| Date: 15 <sup>th</sup> Decembe | er, 2014 | | | | |
|---|---|---|---|---|---|
| Article Title: | | | | | |
| COMPARATIVE | CLINICAL | EVALUATION | OF | SEMILUNAR | CORONALLY |
| POSITIONED FLAP ALONE AND SEMILUNAR CORONALLY POSITIONED FLAP IN | | | | | |
| CONJUNCTION WITH FREE GINGIVAL GRAFT FOR ROOT COVERAGE. | | | | | |
| NCT number: NCT03370042 | | | | | |
| CONSENT | | | | | |
| Ι, | | aged ye | ars h | ave been expl | ained about my |
| participation in the study conducted by Dr. J. Raga Bindu. I am willing for any Photographs | | | | | |
| to be taken, surgical procedure to be carried out and any medication to be prescribed. | | | | | |
| I am willing to do such procedure by my own free will in my conscious presence of mind and | | | | | |
| senses, contributing towards the same after understanding the procedure in my vernacular | | | | | |
| language. | | | | | |
| Date | | | | | |
| | | | | Si | gnature of Patient |